CLINICAL TRIAL: NCT06745570
Title: Improving Sleep As a Method for Enhancing Decision-Making and Reducing Problematic Eating Behaviors in Adolescents with Obesity
Brief Title: Improving Sleep, Decision-Making, and Eating in Adolescents with Obesity
Acronym: STAR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Stephanie Manasse, Assistant Professor, Drexel University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2310010117; R03DK138216 (NIH)
Record Dates: First submitted 2024-12-09; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Adolescent Overweight; Adolescent Obesity; Sleep; Eating Behaviors; Dietary Intake
Keywords: Adolescent Weight Loss; Adolescent Sleep; Adolescent Eating
MeSH Terms: conditions — Pediatric Obesity; Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Group Intervention (Experimental): All participants will receive group-based lifestyle modification and sleep treatment (16, 90-minute sessions over 16 weeks). All sessions will be delivered on Zoom (remotely) to small groups (n=5-10 each) of participants. The intervention involves lifestyle modification content (e.g., nutritional education, physical activity education, stimulus control, goal setting) and sleep content (e.g., psychoeducation regarding sleep and eating behavior, sleep tracking, establishing regular sleep-wake times).
  Interventions: Behavioral: Lifestyle Modification and Sleep Intervention

INTERVENTIONS:
Behavioral: Lifestyle Modification and Sleep Intervention — This study is being performed to develop, refine, and test the effects of a group lifestyle modification intervention augmented with a sleep intervention on weight loss, eating behaviors, and sleep outcomes. Results from this study will inform future studies to test the efficacy of this intervention. This intervention is being offered as part of a research study within Drexel University's WELL Center. Participants will receive remote, group-based, weekly weight loss and sleep coaching (90 minutes per coaching session) for 16 weeks.

SUMMARY:
This study is being performed to understand the effects of a lifestyle modification and sleep intervention on weight loss outcomes in adolescence. The main question the study aims to answer is:

- What are the initial effects of a lifestyle modification and sleep intervention, including effects on weight, eating behaviors and dietary intake, and sleep?

Participants will:

* Participate in remote, group-based, weekly weight loss and sleep coaching for 16 weeks.
* Complete study assessments at baseline (pre-intervention), mid-intervention, and post-intervention.
* Complete daily sleep diaries for three 7-day periods at each assessment point.

DETAILED DESCRIPTION:
In this study, the investigators will develop, refine, and test a 16-session group-based lifestyle modification intervention for adolescents with overweight and obesity augmented with a sleep intervention. The investigators will develop the manual and pilot the intervention in an initial set of adolescents (n=10). The investigators will collect feedback from adolescents, parents, and clinicians, which will inform manual refinements. The investigators will complete an open trial (n=40) of the refined manual. For both phases, the investigators will recruit adolescents (ages 14-18) with overweight or obesity who endorse at least 1 type of sleep disturbance (i.e., too little, poor quality, poorly timed, or inconsistent sleep). Assessments of sleep, decision-making, problematic eating behaviors, energy intake, and weight will occur at baseline (week 0), mid-intervention (week 8) and post-intervention (week 16).

ELIGIBILITY:
Inclusion Criteria:

* Ages 14-18
* Fluent in English
* BMI percentile ≥ 85th percentile for sex-and-age
* Has a parent or guardian who is willing and able to participate
* Has at least one sleep disturbance. Eligible sleep disturbances are: a. Advanced sleep timing (sleep onset 11:00pm or later for 14-16 year-olds or 11:20pm or later for 17-18 year-olds at least 3 times per week), b. Difficulty falling asleep (taking ≥ 30 mins to get to sleep 3 or more nights per week), c. Short sleep (obtaining < 7.5 hours of sleep per night 3 or more nights per week), and d. Sleep irregularity (having more than 2 hours of variability in sleep-wake schedule across one week

Exclusion Criteria:

* Experience of weight loss of ≥ 5% of body weight in the past 6 months
* Current use of insomnia medication
* Having recently begun or changed the dosage of any medication known to affect appetite or body composition within the last 3 months
* Currently taking weight loss medications
* Currently taking insulin
* Diagnosed diabetes (type 1)
* Any condition prohibiting physical activity
* Diagnosis of an eating disorder
* Diagnosis of obstructive sleep apnea
* Recent or ongoing problem with drug abuse, alcohol abuse, or addiction
* Currently pregnant or less than 3 months postpartum
* Anticipation of a possible pregnancy in the next year
* Unwillingness to report possible or confirmed pregnancies promptly during the course of the trial
* Currently participating in treatment for eating or weight concerns
* Does not have regular access to Wi-Fi connection to participate in study interventions.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04-18 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Percent of 95th percentile BMI | From enrollment to the end of the study (approximately 4 months)
  Height and weight will be measured at each assessment and used to calculate percent of 95th percentile BMI.
Tri-ponderal mass index | From enrollment to the end of the study (approximately 4 months)
  The investigators will also calculate tri-ponderal mass index (TMI; i.e., mass divided by height cubed) from measurements of height and weight.
Body fat percentage | From enrollment to the end of the study (approximately 4 months)
  Body fat percentage will also be derived from the Aria Air scale.

SECONDARY OUTCOMES:
Dietary intake | From enrollment to the end of the study (approximately 4 months)
  Adolescent dietary intake will be assessed via 30-day dietary recalls using the VioScreen at the baseline and post-treatment assessments. This freely available and validated web-based tool enables automated, self-administered, 30-day recalls. The VioScreen provides item-level nutritional information as well as monthly totals of key nutrient variables. Mean intake of the following food/macronutrient groups will be calculated: fruits and vegetables, fat, saturated fat, protein, cholesterol, added sugars, and dietary fiber.
Eating Disorder Examination | From enrollment to the end of the study (approximately 4 months)
  The investigators will also assess adolescent eating behaviors using the Binge Module and the Compensatory Behaviors Module portions of the Eating Disorder Examination at each assessment point.
Eating Disorder Examination Questionnaire | From enrollment to the end of the study (approximately 4 months)
  The investigators will have adolescents and their parents complete the Eating Disorder Examination Questionnaire, a self-report measure of eating behaviors, and baseline and post-treatment.
Average total sleep time | From enrollment to the end of the study (approximately 4 months)
  Adolescent sleep diaries will be collected for a 1-week period prior to the initiation of the intervention, 1 week at mid-intervention and 1 week following the intervention. Average total sleep time will be calculated.
Average bed time | From enrollment to the end of the study (approximately 4 months)
  Adolescent sleep diaries will be collected for a 1-week period prior to the initiation of the intervention, 1 week at mid-intervention and 1 week following the intervention. Average bed time will be calculated.
Average sleep latency | From enrollment to the end of the study (approximately 4 months)
  Adolescent sleep diaries will be collected for a 1-week period prior to the initiation of the intervention, 1 week at mid-intervention and 1 week following the intervention. Average sleep latency will be calculated.
Average weekday-weekend bed time shift | From enrollment to the end of the study (approximately 4 months)
  Adolescent sleep diaries will be collected for a 1-week period prior to the initiation of the intervention, 1 week at mid-intervention and 1 week following the intervention. Average weekday-weekend bed time shift will be calculated.
Pittsburgh Sleep Quality Index | From enrollment to the end of the study (approximately 4 months)
  Adolescents and their parents will complete the Pittsburgh Sleep Quality Index, a well-validated overall measure of sleep quality, at each assessment point.
Morningness Eveningness Questionnaire | From enrollment to the end of the study (approximately 4 months)
  The investigators will use the Morningness Eveningness Questionnaire at each assessment point to assess differences in the degree to which adolescents are active and alert at certain times of the day.
Insomnia Severity Index | From enrollment to the end of the study (approximately 4 months)
  The investigators will have participants complete the Insomnia Severity Index to assess insomnia.
Sleep - Fitbit data | From enrollment to the end of the study (approximately 4 months)
  Participants will wear a FitBit during the assessment weeks, which will gather accelerometry data on sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Manasse, Ph.D., Principal Investigator — Drexel University
Locations (1):
- Drexel University WELL Center, Philadelphia, Pennsylvania, United States